CLINICAL TRIAL: NCT01528839
Title: Supraphysiological Doses of Levothyroxine as Adjunctive Therapy in Bipolar Depression: A Multicenter, Randomized, Double-blind, Placebo-controlled Study.
Brief Title: Supraphysiological Doses of Levothyroxine as Adjunctive Therapy in Bipolar Depression
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Stanley Medical Research Institute (Other)
Responsible Party: Principal Investigator, Thomas Stamm, Associate Director Mood Disorders Research Group Department of Psychiatry and Psychotherapy CCM, Charite University, Berlin, Germany
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1908Si267
Record Dates: First submitted 2012-02-06; First posted 2012-02-08 (Estimated); Last update posted 2012-02-08 (Estimated); Status verified 2012-02

CONDITIONS: Bipolar Disorder
Keywords: Bipolar disorder; Bipolar depression; Thyroid abnormality; mood stabilizer; antidepressants; currently depressed
MeSH Terms: conditions — Bipolar Disorder | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pill (Placebo Comparator)
  Interventions: Drug: Placebo
- L-Thyroxine as addon (Experimental)
  Interventions: Drug: L-Thyroxine

INTERVENTIONS:
Drug: L-Thyroxine — L-Thyroxine as addon to ongoing stable antidepressant and /or mood stabilizing therapy: week 1: 100 mcg; week 2: 200 mcg: week 3 to week 6: 300 mcg
  Arms: L-Thyroxine as addon
Drug: Placebo
  Arms: Pill

SUMMARY:
There is growing evidence that thyroid axis dysfunction may contribute to the pathophysiology of bipolar illness. Open-label studies have consistently demonstrated that the behavioral expression of bipolar disorder can be modified by a change in thyroid status, and in many instances the course of illness is improved through the use of adjunct thyroid hormone treatment. Recent evidence emerged from acute intervention studies that add-on treatment with supraphysiological doses of levothyroxine is an effective augmenting agent in patients with a major depressive episode. The primary goal of this international multicenter trial (5 sites) is to determine in a 13-week, randomized, placebo-controlled design (1 week single-blind placebo run-in, 6 week double-blind, 6 week open-label) the efficacy and safety of add-on treatment with levothyroxine (300 mcg/d) in combination with mood stabilizer/antidepressant therapy in the treatment of patients with bipolar depression. The main hypotheses is: treatment with levothyroxine will result in a significantly greater mean reduction of HRSD total score and in a higher number of responders and remitters compared to placebo treatment. This proposal will build on our pilot data and provide evidence for the use of levothyroxine as an effective augmentation strategy in the treatment of bipolar depression.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of bipolar I or II disorder, currently depressive episode according to the Diagnostic and Statistical Manual of Mental Disorders, Fourth Edition (DSM-IV)
* Hamilton Rating Scale for Depression (HAM-D) 17-item score ≥14, a HAM-D item 1 (depressed mood) score ≥2 at the screening and randomization visits
* Young Mania Rating Scale (YMRS) score ≤12 at the screening and randomization visits.
* Pretreatment with a mood stabilizer and/or an antidepressant at standard doses (Bauer et al. 2007a) for at least six weeks since the last dose adjustment, and for at least two weeks before enrollment
* Serum levels of mood stabilizer were required to be within therapeutic ranges
* TSH levels in normal range (serum TSH 0.3 - 4.7 mU/l)

Exclusion Criteria:

* Any axis I disorder other than bipolar disorder
* Recent ultra-rapid cycling course (12 or more episodes in previous year), - - a diagnosis of substance dependence (DSM-IV) or substance use (except for nicotine) within 12 months before the screening visit
* Clinically significant medical illness, especially severe cardiovascular diseases
* Organic brain disorder
* Current serious suicidal or homicidal risk by clinical judgment of the investigator
* History of previous or current thyroid disease
* Thyroid hormone treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2004-03; Primary Completion 2008-05 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Mean change in Hamilton Rating Scale for Depression (HRSD, 17 items) | baseline and six weeks

SECONDARY OUTCOMES:
Mean change and single items change in the Thyroid Symtom List (TSL) | baseline and six weeks
Remission/Response | six weeks
  Rate of Resonders (>50% decline in HRDS) and Remitters (HRDS- score < 9)after l-Thyroxine addon treatment

CONTACTS AND LOCATIONS:
Locations (5):
- University of California in Los Angeles, Los Angeles, California, United States
- Germany (4):
  - Department of Psychiatry and Psychotherapy, Charité Universitätsmedizin Berlin, Campus Mitte, Berlin, Germany, Berlin
  - Department of Psychiatry, LWL University Hospital, Ruhr University Bochum, Bochum, Germany, Bochum
  - Department of Psychiatry and Psychotherapy, University Hospital Carl Gustav Carus, Technische Universität Dresden, Dresden, Germany, Dresden
  - Department of Psychiatry and Psychotherapy, University of Göttingen, Germany, Göttingen

REFERENCES:
- [Derived] Pilhatsch M, J Stamm T, Stahl P, Lewitzka U, Berghofer A, Sauer C, Gitlin M, Frye MA, Whybrow PC, Bauer M. Treatment of bipolar depression with supraphysiologic doses of levothyroxine: a randomized, placebo-controlled study of comorbid anxiety symptoms. Int J Bipolar Disord. 2019 Oct 4;7(1):21. doi: 10.1186/s40345-019-0155-y. PMID 31583561
- [Derived] Stamm TJ, Lewitzka U, Sauer C, Pilhatsch M, Smolka MN, Koeberle U, Adli M, Ricken R, Scherk H, Frye MA, Juckel G, Assion HJ, Gitlin M, Whybrow PC, Bauer M. Supraphysiologic doses of levothyroxine as adjunctive therapy in bipolar depression: a randomized, double-blind, placebo-controlled study. J Clin Psychiatry. 2014 Feb;75(2):162-8. doi: 10.4088/JCP.12m08305. PMID 24345793